CLINICAL TRIAL: NCT03607851
Title: Efficacy and Safety of Rapid Titration Protocols of Lacosamide: An Exploratory Study
Brief Title: Efficacy and Safety of Rapid Titration Protocols of Lacosamide
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Dongsan Medical Center (Other); Konkuk University (Other)
Responsible Party: Principal Investigator, Sang Kun Lee, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0620181410
Record Dates: First submitted 2018-07-24; First posted 2018-07-31 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Focal Epilepsy
MeSH Terms: conditions — Epilepsies, Partial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional titration group (Active Comparator)
  Interventions: Drug: Lacosamide - conventional titration
- Rapid titration group 1 (Experimental)
  Interventions: Drug: Lacosamide - rapid titration 1
- Rapid titration group 2 (Experimental)
  Interventions: Drug: Lacosamide - rapid titration 2

INTERVENTIONS:
Drug: Lacosamide - conventional titration — Administration of lacosamide by the following schedule, Initial: 50 mg PO BID Increase dose at weekly intervals by 50 mg PO BID; up to 200 mg BID
  Arms: Conventional titration group
Drug: Lacosamide - rapid titration 1 — Administration of lacosamide by the following schedule, Initial: 100 mg PO BID Increase dose to 200 mg BID after one week
  Arms: Rapid titration group 1
Drug: Lacosamide - rapid titration 2 — Administration of lacosamide by the following schedule, Initial: 50 mg PO BID Increase dose every two days by 50 mg PO BID; up to 200 mg BID
  Arms: Rapid titration group 2

SUMMARY:
Three different dose titration schedules are tested to find a way to reduce the titration period of lacosamide

DETAILED DESCRIPTION:
The investigators intend to find a way to reduce the titration period of lacosamide. Dosage of lacosamide is increased from 100-200 mg/d to 400 mg/d by three different titration schedule. Safety of lacosamide administration is primary endpoint. 50% responder rate (seizure reduction) and blood level of lacosamide are investigated for secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-85 years old
* Patients diagnosed with focal epilepsy
* Patients subjected to the addition of lacosamide to treat focal onset seizures according to physician's judgement
* Subjects provided informed consent

Exclusion Criteria:

* Subjects who changed other antiepileptic drugs at the beginning of lacosamide treatment
* Subjects with unstable physical, mental or other disease condition that can impede with accurate evaluation or treatment
* Subjects with terminal illness or general medical condition that can impede with the participation of the clinical trial
* Subjects who do not agree with prior consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2018-08-03 (Actual); Primary Completion 2019-06-07 (Actual); Study Completion 2019-06-07 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | 6 (rapid titration group) or 8 weeks (conventional titration group)
  Number of participants with treatment-related adverse events as assessed by Common Terminology Criteria for Adverse Events (CTCAE) v4.

SECONDARY OUTCOMES:
Reduction of seizure frequency | Baseline, 6 weeks (rapid titration group) or 8 weeks (conventional titration group)
  50% responder rate (percentage of patients achieving a 50% or greater reduction in seizure frequency)
lacosamide drug level in the blood | 2 weeks (rapid titration group) or 4 weeks (conventional titration group)
  lacosamide drug level 1 week after the day of the daily dose of lacosamide reaches 400 mg/day

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Doty P, Hebert D, Mathy FX, Byrnes W, Zackheim J, Simontacchi K. Development of lacosamide for the treatment of partial-onset seizures. Ann N Y Acad Sci. 2013 Jul;1291(1):56-68. doi: 10.1111/nyas.12213. PMID 23859801
- [Background] Ben-Menachem E, Biton V, Jatuzis D, Abou-Khalil B, Doty P, Rudd GD. Efficacy and safety of oral lacosamide as adjunctive therapy in adults with partial-onset seizures. Epilepsia. 2007 Jul;48(7):1308-17. doi: 10.1111/j.1528-1167.2007.01188.x. PMID 17635557
- [Background] Halasz P, Kalviainen R, Mazurkiewicz-Beldzinska M, Rosenow F, Doty P, Hebert D, Sullivan T; SP755 Study Group. Adjunctive lacosamide for partial-onset seizures: Efficacy and safety results from a randomized controlled trial. Epilepsia. 2009 Mar;50(3):443-53. doi: 10.1111/j.1528-1167.2008.01951.x. Epub 2009 Jan 17. PMID 19183227
- [Background] Chung S, Sperling MR, Biton V, Krauss G, Hebert D, Rudd GD, Doty P; SP754 Study Group. Lacosamide as adjunctive therapy for partial-onset seizures: a randomized controlled trial. Epilepsia. 2010 Jun;51(6):958-67. doi: 10.1111/j.1528-1167.2009.02496.x. Epub 2010 Jan 27. PMID 20132285